CLINICAL TRIAL: NCT03185494
Title: Clinical Study of CD19/CD22 Tan CAR T Cells in Relapsed and/or Chemotherapy Refractory B-cell Leukemias and Lymphomas
Brief Title: Treatment of Relapsed and/or Chemotherapy Refractory B-cell Malignancy by Tandem CAR T Cells Targeting CD19 and CD22
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, PI, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-022
Record Dates: First submitted 2017-06-10; First posted 2017-06-14 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2018-07

CONDITIONS: Hematopoietic/Lymphoid Cancer; Adult Acute Lymphoblastic Leukemia in Remission; B-cell Adult Acute Lymphoblastic Leukemia; B-Cell Chronic Lymphocytic Leukemia in Relapse (Diagnosis); Prolymphocytic Leukemia; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Refractory Chronic Lymphocytic Leukemia; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Disease; Leukemia, Prolymphocytic; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19/22 CAR T cells (Experimental): Patients receive anti-CD19/22-CAR retroviral vector-transduced autologous or donor-derived T cells on days 0,1, 2 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: anti-CD19/22-CAR vector-transduced T cells

INTERVENTIONS:
Biological: anti-CD19/22-CAR vector-transduced T cells — genetically engineered lymphocyte therapy
  Other Names: genetically engineered lymphocyte therapy

SUMMARY:
RATIONALE: Placing a tumor antigen chimeric receptor that has been created in the laboratory into patient autologous or donor-derived T cells may make the body build immune response to kill cancer cells.

PURPOSE: This clinical trial is studying genetically engineered lymphocyte therapy in treating patients with B-cell leukemia or lymphoma that is relapsed (after stem cell transplantation or intensive chemotherapy) or refractory to chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and feasibility of the chimeric antigen receptor T cells transduced with the anti-CD19/CD22 vector (referred to as tanCART-19/22 cells).

II. Determine duration of in vivo survival of tanCART-19/22 cells. RT-PCR (reverse transcription polymerase chain reaction) analysis of whole blood will be used to detect and quantify survival of tanCART-19/22TCR (T-cell receptor) zeta:CD137 and TCR zeta cells over time.

SECONDARY OBJECTIVES:

I. For patients with detectable disease, measure anti-tumor response due to tanCART-19/22 cell infusions.

II. CD137 transgene is measured by the relative engraftment levels of tanCART-19/22 CD137 and TCR zeta cells over time.

III. Estimate relative trafficking of tanCART-19/22 cells to tumor in bone marrow and lymph nodes.

IV. For patients with stored or accessible tumor cells (such as patients with active chronic lymphocytic leukemia(CLL), acute lymphocytic leukemia (ALL), etc) determine tumor cell killing by tanCART-19/22 cells in vitro.

V. Determine if cellular or humoral host immunity develops against the murine anti-CD19/22, and assess correlation with loss of detectable tanCART-19/20 (loss of engraftment).

VI. Determine the relative subsets of tanCART-19/22 T cells (Tcm, Tem, and Treg).

OUTLINE: Patients are assigned to 1 group according to order of enrollment. Patients receive anti-CD19/22-CAR (coupled with CD137 and CD3 zeta signalling domains)vector-transduced autologous T cells on days 0,1, and 2 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed intensively for 6 months, every 3 months for 2 years, and annually thereafter for 13 years.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with CD19/22+ B cell malignancies in patients with no available curative treatment options (such as autologous or allogeneic SCT) who have limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled CD19/22+ leukemia or lymphoma ALL in CR2(second complete remission) or CR3(third complete remission) and not eligible for allogeneic SCT because of age, comorbid disease, or lack of available family member or unrelated donor

Follicular lymphoma, previously identified as CD19/22+:

At least 2 prior combination chemotherapy regimens (not including single agent monoclonal antibody (Rituxan) therapy Stage III-IV disease Less than 1 year between last chemotherapy and progression (i.e. most recent progression free interval < 1 year) Disease responding or stable after most recent therapy (chemotherapy, MoAb, etc)

CLL:

At least 2 prior chemotherapy regimens (not including single agent monoclonal antibody (Rituxan) therapy. Patients with high risk disease manifested by deletion chromosome 17p will be eligible if they fail to achieve a CR to initial therapy or progress within 2 years of 1 prior Less than 2 years between last chemotherapy and progression (i.e. most recent progression free interval < 2 years) Not eligible or appropriate for conventional allogeneic SCT Patients who achieve only a partial response to FCR(fludarabine, cyclophosphamide and Rituxan) as initial therapy will be eligible.

Mantle cell lymphoma:

Beyond 1st CR (complete remission) with relapsed or persistent disease and not eligible or appropriate for conventional allogeneic or autologous SCT Disease responding or stable after most recent therapy (chemotherapy, MoAb, etc...) Relapsed after prior autologous SCT B-cell prolymphocytic leukemia (PLL) with relapsed or residual disease after at least 1 prior therapy and not eligible for allogeneic SCT

Diffuse large cell lymphoma, previously identified as CD19+:

Residual disease after primary therapy and not eligible for autologous SCT Relapsed after prior autologous SCT Beyond 1st CR with relapsed or persistent disease and not eligible or appropriate of conventional allogeneic or autologous SCT Expected survival > 12 weeks Creatinine < 2.5 mg/dl ALT(alanine aminotransferase)/AST (aspartate aminotransferase)< 3x normal Bilirubin < 2.0 mg/dl Any relapse after prior autologous SCT will make patient eligible regardless of other prior therapy Adequate venous access for apheresis, and no other contraindications for leukapheresis Voluntary informed consent is given

Exclusion Criteria:

* Pregnant or lactating women The safety of this therapy on unborn children is not known Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion Uncontrolled active infection Active hepatitis B or hepatitis C infection Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary Previously treatment with any gene therapy products Feasibility assessment during screening demonstrates < 30% transduction of target lymphocytes, or insufficient expansion (< 5-fold) in response to CD3/CD137 costimulation Any uncontrolled active medical disorder that would preclude participation as outlined HIV infection

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | Until week 24
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment

SECONDARY OUTCOMES:
Anti-tumor responses to tanCART19/22 cell infusions | up to 24 weeks

OTHER OUTCOMES:
in vivo existence of tanCART19/22 | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department and Pediatrics Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Dai H, Wu Z, Jia H, Tong C, Guo Y, Ti D, Han X, Liu Y, Zhang W, Wang C, Zhang Y, Chen M, Yang Q, Wang Y, Han W. Bispecific CAR-T cells targeting both CD19 and CD22 for therapy of adults with relapsed or refractory B cell acute lymphoblastic leukemia. J Hematol Oncol. 2020 Apr 3;13(1):30. doi: 10.1186/s13045-020-00856-8. PMID 32245502